CLINICAL TRIAL: NCT02648217
Title: A Trial Comparing Efficacy and Safety of Insulin Degludec/Insulin Aspart Twice Daily and Biphasic Insulin Aspart Twice Daily in Subjects With Type 2 Diabetes Mellitus Before, During and After Ramadan
Brief Title: Comparing Efficacy and Safety of Insulin Degludec/Insulin Aspart Twice Daily and Biphasic Insulin Aspart Twice Daily in Subjects With Type 2 Diabetes Mellitus Before, During and After Ramadan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-4243; U1111-1170-8304 (Other: WHO)
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2017-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp U100 BID (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- BIAsp U100 BID (Active Comparator)
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Injected subcutaneously (s.c., under the skin)twice daily. The pre-trial insulin will be discontinued.
  Arms: IDegAsp U100 BID
Drug: biphasic insulin aspart — Injected subcutaneously (s.c., under the skin)twice daily. The pre-trial insulin will be discontinued.
  Arms: BIAsp U100 BID

SUMMARY:
This trial is conducted in Africa and Asia. The aim of this trial is to compare efficacy and safety of insulin degludec/insulin aspart twice daily and biphasic insulin aspart twice daily in subjects with type 2 diabetes mellitus before, during and after Ramadan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years at the time of signing informed consent. Algeria: Male or female, age at least 19 years at the time of signing informed consent
* Subjects diagnosed (clinically) with type 2 diabetes mellitus prior to day of screening (Visit 1)
* Treated with any pre-mix/self-mix or basal insulin regimen for at least 90 days prior to the day of screening (Visit 1)
* Subjects not on any OAD(s) (oral anti-diabetic drug) prior to trial participation OR subjects on fixed daily dose(s) of OAD(s) for at least 90 days prior to screening (Visit 1). The OAD(s) include any of the following anti-diabetic drug(s)/regimen: Biguanides (metformin equal to or above 1500 mg or maximum tolerated dose documented in the subject medical record) Insulin secretagogues (sulfonylureas (SU) and glinides), Dipeptidyl peptidase-4 inhibitors (DPP-4 inhibitors), a-glucosidase inhibitors, Sodium-glucose co-transporter 2- inhibitors (SGLT2 Inhibitors ) (above or equal to half of the maximum approved dose according to local label or maximum tolerated dose as documented in subject medical record)
* HbA1c 7.0%-10.0% (53-86 mmol/mol) (both inclusive, by central laboratory analysis)
* Intention to fast (daytime, i.e., between dawn and sunset) during Ramadan after receiving medical counselling regarding the risk of fasting
* Willing to give blood during Ramadan

Exclusion Criteria:

* Any contraindication for successful and sustained fasting from a medical perspective at the discretion of the investigator (such as acute illness, severe hypoglycaemia within 90 days prior to screening (Visit 1), hypoglycaemia unawareness, ketoacidosis within 90 days prior to screening (Visit), hyperosmolar hyperglycaemic coma within 90 days prior to screening (Visit 1), subjects performing intense physical labour)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-09-04 (Actual); Study Completion 2016-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (26):
- Algeria (4):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Sétif
  - Novo Nordisk Investigational Site, Sidi Bel Abbes
- India (7):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Mysore, Karnataka
  - Novo Nordisk Investigational Site, Kozhikode, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
- Lebanon (3):
  - Novo Nordisk Investigational Site, Beirut
  - Novo Nordisk Investigational Site, Hazmiyeh
  - Novo Nordisk Investigational Site, Lebanon - Beirut
- Malaysia (3):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Seremban, Negeri Sembilan
- South Africa (6):
  - Novo Nordisk Investigational Site, Benoni, Gauteng
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Lenasia, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- United Arab Emirates (3):
  - Novo Nordisk Investigational Site, Ajman
  - Novo Nordisk Investigational Site, Dubai
  - Novo Nordisk Investigational Site, Umm Al Quwain City

REFERENCES:
- [Result] Hassanein M, Echtay AS, Malek R, Omar M, Shaikh SS, Ekelund M, Kaplan K, Kamaruddin NA. Original paper: Efficacy and safety analysis of insulin degludec/insulin aspart compared with biphasic insulin aspart 30: A phase 3, multicentre, international, open-label, randomised, treat-to-target trial in patients with type 2 diabetes fasting during Ramadan. Diabetes Res Clin Pract. 2018 Jan;135:218-226. doi: 10.1016/j.diabres.2017.11.027. Epub 2017 Nov 26. PMID 29183844
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 27 sites in 5 countries as follows: Algeria: 4 sites; India: 7 sites; Lebanon: 4 sites; Malaysia: 3 sites; South Africa: 9 sites.
Groups:
- Insulin Degludec/Insulin Aspart: Subjects received insulin degludec/insulin aspart (IDegAsp) subcutaneously (s.c.; under the skin) in the thigh, upper arm or abdomen for a duration of 16-28 weeks (8-20 weeks treatment initiation period [pre-Ramadan], 4-week Ramadan treatment period, and 4 week post-Ramadan period). IDegAsp was administered twice daily (BID) during the entire treatment period with the breakfast/lunch meal and evening meal (during Ramadan Suhur and Iftar), with or without OADs. Subjects on pre-trial basal, premixed or self-mixed insulin therapy were converted unit-to-unit to trial insulin, BID IDegAsp at the same total insulin dose as the subject's pre-trial total daily insulin dose. Subjects used a fixed dose adjustment titration algorithm and there was no minimum or maximum dose for trial products. To optimise and maintain glycaemic control, IDegAsp dose was adjusted based on the subjects' SMPG values, measured twice daily during pre-Ramadan and post-Ramadan and 4 times daily during Ramadan.
- Biphasic Insulin Aspart 30: Subjects received biphasic insulin aspart 30 (BIAsp 30) s.c. in the thigh, upper arm or abdomen for a duration of 16-28 weeks (8-20 weeks treatment initiation period [pre-Ramadan], 4-week Ramadan treatment period, and 4 week post-Ramadan period). BIAsp 30 was administered BID during the entire treatment period with the breakfast/lunch meal and evening meal (during Ramadan Suhur and Iftar), with or without oral antidiabetic drugs (OADs). Subjects on pre-trial basal, premixed or self-mixed insulin therapy were converted unit-to-unit to trial insulin, BID BIAsp 30 at the same total insulin dose as the subject's pre-trial total daily insulin dose. Subjects used a fixed dose adjustment titration algorithm and there was no minimum or maximum dose for trial products. To optimise and maintain glycaemic control, BIAsp 30 dose was adjusted based on the subjects' self-measured plasma glucose (SMPG) values, measured twice daily during pre-Ramadan and post-Ramadan, and 4 times daily during Ramadan
Period: Overall Study
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Started | 131 | 132
Exposed | 130 | 132
Completed | 121 | 127
Not Completed | 10 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Unclassified | 5 | 0

BASELINE CHARACTERISTICS:
Population: Baseline results are based on the full analysis set (FAS), which included all randomised subjects.
Groups:
- Insulin Degludec/Insulin Aspart: Subjects received IDegAsp s.c. in the thigh, upper arm or abdomen for a duration of 16-28 weeks (8-20 weeks treatment initiation period [pre-Ramadan], 4-week Ramadan treatment period, and 4 week post-Ramadan period). IDegAsp was administered BID during the entire treatment period with the breakfast/lunch meal and evening meal (during Ramadan Suhur and Iftar), with or without OADs. Subjects on pre-trial basal, premixed or self-mixed insulin therapy were converted unit-to-unit to trial insulin, BID IDegAsp at the same total insulin dose as the subject's pre-trial total daily insulin dose. Subjects used a fixed dose adjustment titration algorithm and there was no minimum or maximum dose for trial products. To optimise and maintain glycaemic control, IDegAsp dose was adjusted based on the subjects' SMPG values, measured twice daily during pre-Ramadan and post-Ramadan and 4 times daily during Ramadan.
- Biphasic Insulin Aspart 30: Subjects received BIAsp 30 s.c. in the thigh, upper arm or abdomen for a duration of 16-28 weeks (8-20 weeks treatment initiation period [pre-Ramadan], 4-week Ramadan treatment period, and 4 week post-Ramadan period). BIAsp 30 was administered BID during the entire treatment period with the breakfast/lunch meal and evening meal (during Ramadan Suhur and Iftar), with or without OADs. Subjects on pre-trial basal, premixed or self-mixed insulin therapy were converted unit-to-unit to trial insulin, BID BIAsp 30 at the same total insulin dose as the subject's pre-trial total daily insulin dose. Subjects used a fixed dose adjustment titration algorithm and there was no minimum or maximum dose for trial products. To optimise and maintain glycaemic control, BIAsp 30 dose was adjusted based on the subjects' SMPG values, measured twice daily during pre-Ramadan and post-Ramadan, and 4 times daily during Ramadan.
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30 | Total
Number analyzed (Participants) | 131 | 132 | 263
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (9.8) | 55.3 (9.2) | 55.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 80 | 147
  Male | 64 | 52 | 116
Glycated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.5 (0.9) | 8.5 (0.9) | 8.5 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — Population: The number of subjects analysed specifies the number of subjects who contributed to the analysis.
  mmol/L
    number analyzed (Participants) | 124 | 122 | 246
    (all) | 9.9 (10.4) | 10.6 (16.3) | 10.3 (13.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (%) (Glycosylated Haemoglobin)
Description: Mean change in HbA1c was evaluated from baseline (week 0) to end of Ramadan (day 29 of Ramadan).
Time Frame: From week 0 to end of Ramadan (day 29 of Ramadan)
Population: Here, 'number of subjects analysed' specifies the number of subjects, who contributed to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%) of HbA1c
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Number analyzed (Participants) | 121 | 124
Percentage (%) of HbA1c | -1.11 (0.13) | -1.13 (0.13)
Statistical Analysis 1: Comparison: Insulin Degludec/Insulin Aspart vs Biphasic Insulin Aspart 30; The endpoint was analysed using mixed model for repeated measurements (MMRM) with an unstructured covariance matrix. The model included treatment, sex, region, previous OAD treatment, pre-Ramadan trial exposure and visit as factors and age and baseline value of the endpoint as covariates. Interactions between visit and all factors and covariates are included in the model; Test type: Superiority or Other; p = 0.8426, Mixed model for repeated measurements; Treatment Contrast = 0.02, 95% CI 2-sided [-0.20 to 0.24]

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Mean change in FPG was evaluated from baseline (week 0) to end of Ramadan (day 29 of Ramadan).
Time Frame: From week 0 to end of Ramadan (day 29 of Ramadan)
Population: Analysis was based on the FAS, which included all randomised subjects. Here, 'number of subjects analysed' specifies the number of subjects with available data at specified time-point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Number analyzed (Participants) | 115 | 113
mmol/L | -2.0 (12.4) | -4.4 (18.0)

3. Secondary Outcome: Change in Fructosamine
Description: Mean change in fructosamine was evaluated from baseline (week 0) to end of Ramadan (day 29 of Ramadan).
Time Frame: From week 0 to end of Ramadan (day 29 of Ramadan)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Number analyzed (Participants) | 118 | 119
mmol/L | -0.035 (0.051) | -0.035 (0.048)

4. Secondary Outcome: Number of Subjects Who Achieve HbA1c Below 7% (53 mmol/Mol (American Diabetes Association (ADA) Target )
Description: Number of subjects who achieved HbA1c below 7% (53 mmol/mol; ADA target) at the end of Ramadan (day 29 of Ramadan).
Time Frame: End of Ramadan (day 29 of Ramadan)
Population: as for outcome 2
Measure: Number; unit: Number of subjects
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Number analyzed (Participants) | 121 | 123
Number of subjects
  Subjects with HbA1c <7.0% (Yes) | 38 | 42
  Subjects with HbA1c <7.0% (No) | 83 | 81

5. Secondary Outcome: Number of Subjects Who Achieve FPG Below or Equal to 7.2 mmol/L (ADA Target)
Description: Number of subjects who achieved FPG <=7.2 mmol/L at the end of Ramadan (day 29 of Ramadan). The above written (in the endpoint title) 'ADA target' is not applicable for FPG.
Time Frame: End of Ramadan (day 29 of Ramadan)
Population: as for outcome 2
Measure: Number; unit: Number of subjects.
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Number analyzed (Participants) | 121 | 123
Number of subjects.
  Subjects with FPG <=7.2 mmol/L (Yes) | 65 | 83
  Subjects with FPG <=7.2 mmol/L (No) | 56 | 40

6. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Both According to the Novo Nordisk Definition for Hypoglycaemic Episodes (Severe or BG Hypoglycaemia) as Well as According to the ADA definition1 Confirmed Symptomatic
Description: Treatment-emergent hypoglycaemic episodes: If the onset of the episode occurred on or after the first day of investigational medicinal product (IMP; IDegAsp/BIAsp 30) administration, and no later than 1 day after the last day on IMP, before switching to or being treated with another insulin product.
  The above mentioned definitions (in endpoint title) should read as the following:
  Novo Nordisk definition; severe or blood glucose (BG) confirmed symptomatic hypoglycaemia: An episode that was severe according to ADA classification or BG confirmed by a plasma glucose (PG) value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  American Diabetes Association (ADA) definition; documented symptomatic hypoglycaemia: An episode, during which typical symptoms of hypoglycaemia were accompanied by a measured PG concentration ≤3.9 mmol/L (70 mg/dL).
  Due to character limitation, severe hypoglycaemia as per ADA classification is not defined here; see next outcome measure.
Time Frame: From week 0 to 4 weeks post Ramadan
Population: Analysis was based on the safety analysis set (SAS), which included all subjects receiving at least 1 dose of the investigational product (IDegAsp) or its comparator (BIAsp 30).
Measure: Number; unit: Number of episodes.
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Number analyzed (Participants) | 130 | 132
Number of episodes.
  Severe or BG confirmed symptomatic hypoglycaemia | 93 | 389
  Documented symptomatic hypoglycaemia | 521 | 775

7. Secondary Outcome: Number of Treatment Emergent Nocturnal (00:01-05:59 am) Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes, which occurred between 00:01 and 05:59 both inclusive.
  Novo Nordisk definition; severe or blood glucose (BG) confirmed symptomatic hypoglycaemia: An episode that was severe according to ADA classification or BG confirmed by a plasma glucose (PG) value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  Severe hypoglycaemia as per ADA classification: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: From week 0 to 4 weeks post Ramadan
Population: Analysis was based on the SAS, which included all subjects receiving at least one dose of the investigational product or its comparator.
Measure: Number; unit: Number of episodes.
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Number analyzed (Participants) | 130 | 132
Number of episodes. | 18 | 106

ADVERSE EVENTS:
Time Frame: From first day of exposure to randomised treatment (week 0) and no later than seven days after the last day of randomised treatment (i.e., after 16-28 weeks; 8-20 weeks treatment initiation period [pre-Ramadan], 4-week Ramadan treatment period, and 4 week post-Ramadan period).
Description: All the adverse events mentioned below are treatment-emergent. A treatment-emergent adverse event (TEAE) was defined as an event that had an onset date on or after the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment. Analysis was based on the SAS, which included all subjects receiving at least one dose of the investigational product or its comparator.
Arm/Group | Insulin Degludec/Insulin Aspart | Biphasic Insulin Aspart 30
Serious Adverse Events (participants affected / at risk) | 5/130 | 3/132
Other Adverse Events (participants affected / at risk) | 54/130 | 47/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Insulin Aspart (N=130) | Biphasic Insulin Aspart 30 (N=132)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (7)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Insulin Aspart (N=130) | Biphasic Insulin Aspart 30 (N=132)
Blood glucose decreased (Investigations) | 46 (115) | 40 (89)
Pyrexia (General disorders) | 4 (4) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.